CLINICAL TRIAL: NCT05330130
Title: Impact of FSH Dosage During Ovarian Stimulation for IVF/ICSI on the Expression of FSH- and LH-receptors in Granulosa Cells
Brief Title: Impact of FSH Dosage During Ovarian Stimulation for IVF/ICSI in Granulosa Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Collaborators: Organon and Co (Industry)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2107-ABU-010-BL
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Function Insufficiency; Fertility Issues; Infertility,Female; Infertility
Keywords: Ovarian stimulation; Granulosa cells; Follicle Stimulating Hormone Receptor; Luteinising Hormone Receptor; Elevated progesterone
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — follitropin beta; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily 150 IU recFSH (Active Comparator): Follitropin beta injection 150 IU daily
  Interventions: Drug: Follitropin beta injection 150 IU
- Daily 300 IU recFSH (Active Comparator): Follitropin beta injection 300 IU daily
  Interventions: Drug: Follitropin beta injection 300 IU

INTERVENTIONS:
Drug: Follitropin beta injection 150 IU — Participants commence ovarian stimulation on day 2 or 3 of their menstrual cycle with a daily dosage of 150 IU rec-FSH. The dosage will remain constant throughout the course of the stimulation. From the morning of the 5th stimulation day, GnRH-antagonist will be administered daily to prevent LH-rise. As soon as ≥ 3 follicle of a size of 17mm are seen, 0.3 mg GnRH-Agonist will be administered for final oocyte maturation. During ovarian stimulation, follicle puncture procedures with the aspiration of follicular fluid will be performed at the following time:
  * one follicle on the morning of day 5, before the administration of the first GnRH-antagonist
  * one follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm
  * two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation.
  Oocyte retrieval of all other follicles will be carried out 36 hours after injection of the medication for final oocyte maturation.
  Other Names: FOLLISTIM AQ
  Arms: Daily 150 IU recFSH
Drug: Follitropin beta injection 300 IU — Participants commence ovarian stimulation on day 2 or 3 of their menstrual cycle with a daily dosage of 300 IU rec-FSH. The dosage will remain constant throughout the course of the stimulation. From the morning of the 5th stimulation day, GnRH-antagonist will be administered daily to prevent LH-rise. As soon as ≥ 3 follicle of a size of 17mm are seen, 0.3 mg GnRH-Agonist will be administered for final oocyte maturation. During ovarian stimulation, follicle puncture procedures with the aspiration of follicular fluid will be performed at the following time:
  * one follicle on the morning of day 5, before the administration of the first GnRH-antagonist
  * one follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm
  * two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation.
  Oocyte retrieval of all other follicles will be carried out 36 hours after injection of the medication for final oocyte maturation.
  Other Names: FOLLISTIM AQ
  Arms: Daily 300 IU recFSH

SUMMARY:
To study the influence of different daily rec-FSH dosages (150 IU versus 300 IU), performed in the same patient in consecutive cycles, on the relation between FSH- and LH-receptors of the granulosa cells of the growing follicle.

DETAILED DESCRIPTION:
This is a prospective cross-over study. Investigators want to study the effect of different dosages of recombinant FSH in the same patient on the expression of the FSH- and LH-receptors in the granulosa cells and on the endocrine milieu in the blood and the follicular fluid. An improved understanding of the mechanism leading to progesterone elevation might initiate a change in the ovarian stimulation approach, thereby not only preventing progesterone elevation and its negative consequences on ART (Assisted Reproductive Technology) outcome, but also improving individualization of the ovarian stimulation treatment according to the patients' characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Desire to perform oocyte freezing for social fertility preservation, age 18 - 38 years
* BMI of 18-32 kg/m2
* Regular menstrual cycles with a length of 24-35 days
* Anti-Muellerian-Hormone levels between 1.3 - 6.25 ng/ml (Ferraretti and Gianaroli, 2014; Calzada et al., 2019)

Exclusion Criteria:

* Occurrence of ovarian hyperstimulation syndrome (OHSS)
* Occurrence of poor ovarian response (AFC < 5 and AMH < 0,5ng/ml) in previous ovarian stimulation treatment (20)
* Polycystic ovary syndrome (PCOS) (21)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of FSHR- and LHR of the GC, obtained from one follicle on the morning of day 5, before the administration of the first GnRH-antagonist, punctured during the ovarian stimulation cycle | 5 days
Number of FSHR- and LHR of the GC, obtained from tone follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm, punctured during the ovarian stimulation cycle | 1 day
Number of FSHR- and LHR of the GC, obtained from two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation, punctured during the ovarian stimulation cycle | 1 day
Number of FSHR- and LHR of the GC, obtained from the follicular fluid of follicles aspirated during OPU | 1 day

SECONDARY OUTCOMES:
Level of E2 hormone in the blood, the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of P4 hormone in the blood, the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of FSH hormone in the blood, the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of LH hormone in the blood, the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of E2 hormone in the blood, when there are at least 2 to 3 follicles with a size of 12 to 14 mm | 1 day
Level of P4 hormone in the blood, when there are at least 2 to 3 follicles with a size of 12 to 14 mm | 1 day
Level of FSH hormone in the blood, when there are at least 2 to 3 follicles with a size of 12 to 14 mm | 1 day
Level of LH hormone in the blood, when there are at least 2 to 3 follicles with a size of 12 to 14 mm | 1 day
Level of E2 hormone in the blood, on the morning of the day of final oocyte maturation | 1 day
Level of P4 hormone in the blood, on the morning of the day of final oocyte maturation | 1 day
Level of FSH hormone in the blood, on the morning of the day of final oocyte maturation | 1 day
Level of LH hormone in the blood, on the morning of the day of final oocyte maturation | 1 day
Level of E2 hormone in the blood, on the day of OPU | 1 day
Level of P4 hormone in the blood, on the day of OPU | 1 day
Level of FSH hormone in the blood, on the day of OPU | 1 day
Level of LH hormone in the blood, on the day of OPU | 1 day
Level of E2 hormone in the follicular fluid of one follicle on the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of P4 hormone in the follicular fluid of one follicle on the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of FSH hormone in the follicular fluid of one follicle on the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of LH hormone in the follicular fluid of one follicle on the morning of day 5, before the administration of the first GnRH-antagonist | 5 days
Level of E2 hormone in the follicular fluid of one follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm | 1 day
Level of P4 hormone in the follicular fluid of one follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm | 1 day
Level of FSH hormone in the follicular fluid of one follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm | 1 day
Level of LH hormone in the follicular fluid of one follicle of the size of 12 to 14 mm, when at least 2 to 3 follicles have reached a size of 12 to 14 mm | 1 day
Level of E2 hormone in the follicular fluid of two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation | 1 day
Level of P4 hormone in the follicular fluid of two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation | 1 day
Level of FSH hormone in the follicular fluid of two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation | 1 day
Level of LH hormone in the follicular fluid of two follicles (= pre-ovulatory follicle) on the morning of the day of final oocyte maturation | 1 day
Level of E2 hormone in the follicular fluid of follicles aspirated during OPU | 1 day
Level of P4 hormone in the follicular fluid of follicles aspirated during OPU | 1 day
Level of FSH hormone in the follicular fluid of follicles aspirated during OPU | 1 day
Level of LH hormone in the follicular fluid of follicles aspirated during OPU | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker VL, Brown MB, Luke B, Smith GW, Ireland JJ. Gonadotropin dose is negatively correlated with live birth rate: analysis of more than 650,000 assisted reproductive technology cycles. Fertil Steril. 2015 Nov;104(5):1145-52.e1-5. doi: 10.1016/j.fertnstert.2015.07.1151. Epub 2015 Aug 18. PMID 26297646
- [Background] Bosch E, Valencia I, Escudero E, Crespo J, Simon C, Remohi J, Pellicer A. Premature luteinization during gonadotropin-releasing hormone antagonist cycles and its relationship with in vitro fertilization outcome. Fertil Steril. 2003 Dec;80(6):1444-9. doi: 10.1016/j.fertnstert.2003.07.002. PMID 14667881
- [Background] Calzada M, Lopez N, Noguera JA, Mendiola J, Hernandez AI, Corbalan S, Sanchez M, Torres AM. AMH in combination with SHBG for the diagnosis of polycystic ovary syndrome. J Obstet Gynaecol. 2019 Nov;39(8):1130-1136. doi: 10.1080/01443615.2019.1587604. Epub 2019 Jun 17. PMID 31208261
- [Background] Erickson GF, Wang C, Hsueh AJ. FSH induction of functional LH receptors in granulosa cells cultured in a chemically defined medium. Nature. 1979 May 24;279(5711):336-8. doi: 10.1038/279336a0. No abstract available. PMID 221826
- [Background] Fauser BC. Towards the global coverage of a unified registry of IVF outcomes. Reprod Biomed Online. 2019 Feb;38(2):133-137. doi: 10.1016/j.rbmo.2018.12.001. Epub 2018 Dec 14. No abstract available. PMID 30593441
- [Background] Ferraretti AP, Gianaroli L. The Bologna criteria for the definition of poor ovarian responders: is there a need for revision? Hum Reprod. 2014 Sep;29(9):1842-5. doi: 10.1093/humrep/deu139. Epub 2014 Jul 9. PMID 25008235
- [Background] Filicori M, Cognigni GE, Gamberini E, Parmegiani L, Troilo E, Roset B. Efficacy of low-dose human chorionic gonadotropin alone to complete controlled ovarian stimulation. Fertil Steril. 2005 Aug;84(2):394-401. doi: 10.1016/j.fertnstert.2005.02.036. PMID 16084880
- [Background] Huang B, Ren X, Wu L, Zhu L, Xu B, Li Y, Ai J, Jin L. Elevated Progesterone Levels on the Day of Oocyte Maturation May Affect Top Quality Embryo IVF Cycles. PLoS One. 2016 Jan 8;11(1):e0145895. doi: 10.1371/journal.pone.0145895. eCollection 2016. PMID 26745711
- [Background] Jeppesen JV, Kristensen SG, Nielsen ME, Humaidan P, Dal Canto M, Fadini R, Schmidt KT, Ernst E, Yding Andersen C. LH-receptor gene expression in human granulosa and cumulus cells from antral and preovulatory follicles. J Clin Endocrinol Metab. 2012 Aug;97(8):E1524-31. doi: 10.1210/jc.2012-1427. Epub 2012 Jun 1. PMID 22659248
- [Background] Lawrenz B, Beligotti F, Engelmann N, Gates D, Fatemi HM. Impact of gonadotropin type on progesterone elevation during ovarian stimulation in GnRH antagonist cycles. Hum Reprod. 2016 Nov;31(11):2554-2560. doi: 10.1093/humrep/dew213. Epub 2016 Sep 12. PMID 27619773
- [Background] Lawrenz B, Fatemi HM. Effect of progesterone elevation in follicular phase of IVF-cycles on the endometrial receptivity. Reprod Biomed Online. 2017 Apr;34(4):422-428. doi: 10.1016/j.rbmo.2017.01.011. Epub 2017 Jan 24. PMID 28162937
- [Background] Lawrenz B, Labarta E, Fatemi H, Bosch E. Premature progesterone elevation: targets and rescue strategies. Fertil Steril. 2018 Apr;109(4):577-582. doi: 10.1016/j.fertnstert.2018.02.128. PMID 29653703
- [Background] Lawrenz B, Melado L, Fatemi H. Premature progesterone rise in ART-cycles. Reprod Biol. 2018 Mar;18(1):1-4. doi: 10.1016/j.repbio.2018.01.001. Epub 2018 Jan 6. PMID 29317175
- [Background] Macklon NS, Stouffer RL, Giudice LC, Fauser BC. The science behind 25 years of ovarian stimulation for in vitro fertilization. Endocr Rev. 2006 Apr;27(2):170-207. doi: 10.1210/er.2005-0015. Epub 2006 Jan 24. PMID 16434510
- [Background] Munch EM, Sparks AE, Zimmerman MB, Van Voorhis BJ, Duran EH. High FSH dosing is associated with reduced live birth rate in fresh but not subsequent frozen embryo transfers. Hum Reprod. 2017 Jul 1;32(7):1402-1409. doi: 10.1093/humrep/dex094. PMID 28472321
- [Background] Oktem O, Akin N, Bildik G, Yakin K, Alper E, Balaban B, Urman B. FSH Stimulation promotes progesterone synthesis and output from human granulosa cells without luteinization. Hum Reprod. 2017 Mar 1;32(3):643-652. doi: 10.1093/humrep/dex010. PMID 28158500
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Background] Venetis CA, Kolibianakis EM, Bosdou JK, Tarlatzis BC. Progesterone elevation and probability of pregnancy after IVF: a systematic review and meta-analysis of over 60 000 cycles. Hum Reprod Update. 2013 Sep-Oct;19(5):433-57. doi: 10.1093/humupd/dmt014. Epub 2013 Jul 4. PMID 23827986
- [Background] Wilcox AJ, Baird DD, Weinberg CR. Time of implantation of the conceptus and loss of pregnancy. N Engl J Med. 1999 Jun 10;340(23):1796-9. doi: 10.1056/NEJM199906103402304. PMID 10362823
- See also: Segaloff DL, Richards JS, Ascoli M, Wang H. Regulation of the LH/CG Receptor by Gonadotropins. In Hunzicker-Dunn M, Schwartz NB, editors. Follicle Stimul Horm [Internet] 1992;, p. 199-205. Springer New York: New York, NY — http://link.springer.com/10.1007/978-1-4684-7103-8_16